CLINICAL TRIAL: NCT01364896
Title: Characterization of Anal Human Papillomavirus (HPV) Infection in the University of Pittsburgh Inflammatory Bowel Disease (IBD) Cohort Study
Brief Title: Anal Human Papillomavirus in Inflammatory Bowel Disease Study
Acronym: AnalHPV&IBD
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 38458
Record Dates: First submitted 2011-05-26; First posted 2011-06-03 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2016-03

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis (UC); Crohn's Disease (CD); Anal Human Papillomavirus
Keywords: Non-corticosteroid immunosuppressive agent
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood, anal swabs, vaginal swabs, high resolution anoscopy (HRA), anal biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease, Immunosuppressive agent: Men and women 18 years + with a histological diagnosis of IBD (ulcerative colitis or Crohn's disease) who are undergoing a colonoscopy prior to starting a non-corticosteroid immunosuppressive agent
  Interventions: Procedure: Venous blood samples, anal swab samples, vaginal swab samples, high resolution anoscopy (HRA), anal biopsy samples

INTERVENTIONS:
Procedure: Venous blood samples, anal swab samples, vaginal swab samples, high resolution anoscopy (HRA), anal biopsy samples — Before and at least 6 months after starting a new non-steroid immunosuppressive agent for IBD treatment, eligible participants who are attending for routine colonoscopy will have:
  1. Anal swab samples (and vaginal swab samples for female participants) for human papillomavirus PCR typing (6, 11, 16, 18, 31, 33, 45, 52, 58)
  2. High-resolution anoscopy and biopsy of all visible high-grade dysplastic lesions based on validated colposcopic criteria
  3. Anal cytology testing

SUMMARY:
This is an observational cohort study with two time points (baseline and after at least 6 months of treatment with a non-corticosteroid immunosuppressive agent for inflammatory bowel disease (IBD)). Approximately 40 participants, both male and female, 18 years of age and older will be recruited from the Pittsburgh IBD Cohort.

Participants will have a histological diagnosis of IBD (Ulcerative Colitis (UC) or Crohn's Disease (CD)) and will be attending for colonoscopy prior to starting a non-corticosteroid immunosuppressive agent as part of standard medical care. Immediately following the colonoscopy, an anal exam will be performed for research purposes to include:

1. Perianal inspection
2. Anal canal HPV swab
3. Anal cytology
4. Digital anal examination
5. High resolution anoscopy (HRA) and biopsy of all lesions with visual criteria consistent with high-grade anal dysplasia
6. For female participants a self- or clinician-taken vaginal swab for HPV typing.

These procedures will be repeated at routine colonoscopy following at least 6 months but within 12 months of non-corticosteroid immunosuppressive treatment.

DETAILED DESCRIPTION:
Treatment of IBD relies on disease modification by induction of relative immunosuppression with corticosteroids and latterly and increasingly, by the use of immunomodulators (azathioprine, mercaptopurine, methotrexate), biological agents such as anti tumor necrosis factor monoclonal antibodies (infliximab, adalimumab, certolizumab) or with a circulating receptor fusion protein (etanercept). These agents impair cell mediated immunity (CMI) and have been associated with increased rates of both tuberculosis and fungal infections in treated populations beyond that seen with corticosteroids alone. Following initial infection, HPV is controlled by CMI and manifestations of infection become increasingly clinically apparent when CMI is impaired due to for example HIV co-infection or systemic immunosuppression. There is appropriate concern in the IBD treatment community that the use of immunosuppression to modify disease course may lead to increased rates of HPV associated disease including warts, dysplasia and ultimately anogenital cancer above and beyond the established increased risk associated with IBD. In this context it is important to establish the prevalence of both HPV infection and anal dysplasia in patients with IBD before and after treatment with a non-steroid immunosuppressive agent. These data will help determine the need for HPV vaccination and/or anal dysplasia screening in patients with IBD.

VISIT 1 (Screening/Enrollment Visit): This visit will include:

* Medical/medication history.
* Physical exam as per standard of care
* Females of reproductive potential will give a urine sample for a pregnancy test. This test must be negative.
* An anal Pap test for abnormal cells. The researcher will insert a swab (similar to a Q-tip) into the anus. The end of the swab will be rubbed against the skin inside the anus.
* An anal swab to test for HPV (using the same method as the anal Pap)
* Female participants will also have a vaginal swab for HPV. This may be self taken, or taken by a clinician.
* An exam of the anus and genital area for any lesions or masses.
* A rectal exam with a finger to feel for any abnormalities.
* An anal exam called high resolution anoscopy (HRA) that uses a special microscope and dyes to examine the anus for abnormal areas. A lubricated plastic speculum will be inserted into the anus. Then, a swab moistened with acetic acid is placed in the anus so that abnormal areas will be visible. A colposcope will be used to view the skin inside the anus. A biopsy, with or without iodine for visualization of the abnormal areas, may be taken if any lesions have the appearance of high-grade anal dysplasia or other abnormal findings.

Within 1 day after this visit, study staff will telephone the participant to ask about any side effects or health problems from the study procedures. If necessary, the participant may be asked to come to the clinic for a visit.

VISIT 2 (Final Visit): This visit will occur 6 to 12 months after the first visit. Prior to this visit, participant will be instructed to not have anal sex or insert anything into the anus, including enemas, for 24 hours before each study visit. This visit will include:

* Medical/medication history
* Physical exam as per standard of care
* Females of reproductive potential will give a urine or 5ml blood sample] for a pregnancy test. This test must be negative.
* Anal Pap test for abnormal cells
* Anal swab for HPV
* Females participants will also have a vaginal swab for HPV
* An exam of the anus and genital area for any lesions, tenderness or masses
* A rectal exam to feel for any abnormalities
* High-resolution anoscopy (HRA). A biopsy, with or without iodine for visualization of the abnormal areas, may be taken if any lesions have the appearance of high-grade anal dysplasia or other abnormal findings.

Within 1 day after this visit, study staff will telephone the participant to ask about any side effects or health problems from the study procedures. If necessary, the participant may be asked to come to the clinic for a visit.

ELIGIBILITY:
Inclusion Criteria:

1. Previous biopsy proven inflammatory bowel disease (ulcerative colitis or Crohn's disease)
2. Male or female over 18 years of age
3. Able and willing to give informed consent in English
4. Able and willing to provide locator information
5. Planned commencement of a non-corticosteroid immunosuppressive agent for management of inflammatory bowel disease
6. Sexually active
7. Female subjects of reproductive potential must agree to use an acceptable method of birth control while on this study.

Exclusion Criteria:

1. Previous or current treatment with a biological agent for inflammatory bowel disease
2. Any other condition or prior therapy that, in the opinion of the investigator, would make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease
3. For female subjects of reproductive potential, current pregnancy, pregnancy within the 90 days prior to study entry, or planning to become pregnant within 12 months after study entry
4. For female subjects, currently breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women 18 years + with a histological diagnosis of IBD (ulcerative colitis or Crohn's disease) who are undergoing a colonoscopy prior to starting a non-corticosteroid immunosuppressive agent
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Cranston, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Inflammatory Bowel Disease, Immunosuppressive Agent: Men and women 18 years + with a histological diagnosis of IBD (ulcerative colitis or Crohn's disease) who are undergoing a colonoscopy prior to starting a non-corticosteroid immunosuppressive agent
  Venous blood samples, anal swab samples, vaginal swab samples, high resolution anoscopy (HRA), anal biopsy samples: Before and at least 6 months after starting a new non-steroid immunosuppressive agent for IBD treatment, eligible participants who are attending for routine colonoscopy will have:
  1. Anal swab samples (and vaginal swab samples for female participants) for human papillomavirus PCR typing (6, 11, 16, 18, 31, 33, 45, 52, 58)
  2. High-resolution anoscopy and biopsy of all visible high-grade dysplastic lesions based on validated colposcopic criteria
  3. Anal cytology testing
Period: Overall Study
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 46
Number of participants with Crohn's Disease [Number; unit: participants] | 31
Number of participants with Ulcerative Colitis [Number; unit: participants] | 14
Number of participants with Indeterminate Colitis [Number; unit: participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anal HPV of Any Type, Single Type, and Multiple Types
Description: Anal (and vaginal for female participants) HPV PCR typing (6, 11, 16, 18, 31, 33, 45, 52, 58) using the SYBR-Green-based real-time PCR assay with a reverse line blot assay for genotyping of HPV in the positive samples and Taqman probe-based real-time PCR assays for quantification of individual HPV subtypes
Time Frame: Baseline and 6 to 12 months
Measure: Number; unit: participants
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 46
participants
  Number of Participants with Anal HPV of Any Type | 41
  Number of Participants with Single Types | 16
  Number of Participants with Multiple Types | 25

2. Primary Outcome: Percent of Participants With HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and/or 58
Time Frame: Baseline and 6 to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 41
percentage of participants
  Percent of Participants with HPV type 6 | 6.6
  Percent of Participants with HPV type 11 | 23.9
  Percent of Participants with HPV type 16 | 65.2
  Percent of Participants with HPV type 18 | 2.2
  Percent of Participants with HPV type 31 | 2.2
  Percent of Participants with HPV type 33 | 0
  Percent of Participants with HPV type 45 | 23.9
  Percent of Participants with HPV type 52 | 0
  Percent of Participants with HPV type 58 | 2.2
  Percent of Females with Vaginal HPV | 90.5

3. Primary Outcome: Number of Participants With Abnormal Anal Cytology (ASC-US, ASC-H, LSIL, HSIL, Cancer)
Description: High-resolution anoscopy with anal cytology testing
Time Frame: Baseline and 6 to 12 months
Measure: Number; unit: participants
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 46
participants
  Number of Participants with Abnormal Anal Cytology | 21
  Number of Participants with Anal Dysplasia | 28
  Number of Participants with HSIL | 4
  Number of Participants with LSIL | 24

4. Primary Outcome: Number of Participants Who Had One or More Anal Biopsies
Description: High resolution anoscopy and biopsy of all visible high-grade dysplastic lesions based on validated colposcopic criteria
Time Frame: Baseline and 6 to 12 months
Measure: Number; unit: participants
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 46
participants | 33

5. Primary Outcome: Number of Participants With High-grade Anal Dysplasia Lesions
Description: as for outcome 4
Time Frame: Baseline and 6 to 12 months
Measure: Number; unit: participants
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Number analyzed (Participants) | 46
participants | 28

ADVERSE EVENTS:
Arm/Group | Inflammatory Bowel Disease, Immunosuppressive Agent
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No